CLINICAL TRIAL: NCT02264834
Title: Comparison of Two Different Peridural During the Labor and Effect of Deambulation
Brief Title: Deambulatory Epidural During the Labour
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr Madeleine Wilwerth (Other)
Responsible Party: Sponsor-Investigator, Dr Madeleine Wilwerth, primary investigator, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PDB001
Record Dates: First submitted 2014-08-01; First posted 2014-10-15 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: First Pregnancy
Keywords: epidural; primiparous patient; deambulation
MeSH Terms: interventions — Levobupivacaine; Sufentanil; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Lumbar epidural analgesia during the labour and end up after delivery Levobupivacaine 0.1% + Sufentanil 0.2 µg/mL
  Interventions: Drug: Levobupivacaine 0.1% + Sufentanil 0.2µg/ml; Procedure: Lumbar epidural analgesia
- Ambulatory group (Experimental): Lumbar epidural analgesia during the labour and end up after delivery Levobupivacaine 0.07% + Sufentanil 0.3 µg/mL
  Interventions: Drug: Levobupivacaine 0.07% + Sufentanil 0.3µg/ml; Procedure: Lumbar epidural analgesia

INTERVENTIONS:
Drug: Levobupivacaine 0.1% + Sufentanil 0.2µg/ml — Levobupivacaine 0.1% + Sufentanil 0.2µg/ml
  Other Names: control group
  Arms: Control group
Drug: Levobupivacaine 0.07% + Sufentanil 0.3µg/ml — Levobupivacaine 0.07% + Sufentanil 0.3µg/ml
  Other Names: ambulatory group
  Arms: Ambulatory group
Procedure: Lumbar epidural analgesia — Introduction of a catheter in lumbar epidural space
  Other Names: labor analgesia

SUMMARY:
Assess the impact of instrumentation and caesarean related to dyskinesia by reducing the concentration of local anesthetic and therefore the motor block.

DETAILED DESCRIPTION:
Prospective, randomized and double-blind study performed on primiparous parturient divided into two distinct groups.

ELIGIBILITY:
Inclusion Criteria:

* Free written consent.
* ASA I or II,
* Primipara, unique and pregnancy over 36 weeks fetus in cephalic, cervical dilation between 3-6 cm
* VAS> 30 mm
* No contraindications to peridural

Exclusion Criteria:

* Twin pregnancy, less than 36 weeks and 42 weeks
* Fetus in breech position
* Analgesia and sedation within 6h
* Contraindications to peridural

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Time between peridural application and childbirth | at delivery
  This will be used to assess labor.
Caesarian | at delivery
  This will be used to assess labor. Was a caesarian necessary (yes-no) ?
Instrumentalisation | at delivery
  This will be used to assess labor. Was an instrumentalisation (defined as the use of forceps or suction cups) necessary at delivery (yes-no) ?
Apgar score of the baby | at delivery
  Evaluation of the baby, using the Apgar score. This will be used to assess labor.

SECONDARY OUTCOMES:
Bromage score | 1h after the start of the peridural
  Modified Bromage score (Breen et al) >5 and ability to stand on one leg alternatively. This will be used to assess perambulation (motricity).
Romberg test | 1h after the start of the peridural
  Romberg test during 20-30 seconds. This will be used to assess perambulation (proprioception).
Arterial tension | 1h after the start of the peridural
  Absence of orthostatic hypotension (i-e less than 20% of the usual arterial tension of the patient).

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Vanderlinden, Study Director — CHUB
Locations (1):
- CHUB, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No